CLINICAL TRIAL: NCT03645902
Title: Comparison Between Enhanced Susceptibility-weighted Angiography and Time of Flight Sequences in the Detection of Arterial Occlusion in Acute Ischemic Stroke Using MRI
Brief Title: Comparison Between TOF and SWAN Sequences in the Detection of Arterial Occlusion in Acute Ischemic Stroke Using MRI
Acronym: TOF-SWAN
Status: Completed | Type: Observational
Sponsor: Lille Catholic University (Other)
Responsible Party: Sponsor
Other Study IDs: TOF-SWAN
Record Dates: First submitted 2018-08-22; First posted 2018-08-24 (Actual); Last update posted 2018-08-24 (Actual); Status verified 2018-08

CONDITIONS: Stroke, Acute; Angiography; Magnetic Resonance Imaging; Diagnosis
Keywords: Acute stroke; Susceptibility-weighted imaging; Arterial occlusion; Time of flight
MeSH Terms: conditions — Stroke; Disease; Arterial Occlusive Diseases | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Acute stroke patients: MRI examinations will be performed on a 3 T GE MR750 W scanner. Two readers, an experienced neuroradiologist (8 years of experience in neuroradiology) and a junior radiologist (3 years of experience in general radiology) will independently analyze eSWAN and TOF images in random order, looking for arterial occlusions. Analysis will be based on a 2-point-scale: arterial occlusion, based on a local signal loss, or acceptable permeability.
  Interventions: Diagnostic Test: Magnetic resonance imaging

INTERVENTIONS:
Diagnostic Test: Magnetic resonance imaging

SUMMARY:
Optimizing the MRI protocol in acute ischemic stroke remains a challenging issue. In this field, susceptibility-weighted sequences have proved their superiority over T2. Besides the strengthened susceptibility effect, enhanced susceptibility-weighted angiography (eSWAN) sequence provides also a time-of-flight (TOF) effect, allowing the exploration of the intracranial arterial circulation. The objective of this study is to compare eSWAN and 3D TOF, considered as the reference, in the detection of arterial occlusion in acute stroke.

DETAILED DESCRIPTION:
Patients who undergo MRI for suspected acute stroke with an acute ischemic lesion on diffusion-weighted imaging (DWI) will be prospectively included in this study.eSWAN and TOF images will be analyzed under double-blind conditions by a junior radiologist and a senior neuroradiologist for the detection of arterial occlusion. eSWAN images will be assessed in order to estimate the inter-observer agreement. After a consensus, eSWAN and TOF data will be compared to calculate inter-modality agreement.

ELIGIBILITY:
Inclusion Criteria:

* clinical symptoms compatible with acute stroke;
* time range between symptoms and magnetic resonance imaging less than 4 h 30
* presence of at least one acute ischemic lesion on the diffusion-weighted images (DWI).

Exclusion Criteria:

* MR contraindications;
* negative DWI;
* differential diagnosis;
* incomplete acquisition of the full magnetic resonance imaging protocol or technical issues leading to uninterpretable eSWAN and/or TOF sequences (e.g.motion artifacts).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients included in this prospective study will be recruited at Saint-Philibert Hospital -Lomme, France, when presenting symptoms of an acute stroke
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2014-03-01 (Actual); Primary Completion 2014-07-31 (Actual); Study Completion 2014-12-31 (Actual)

PRIMARY OUTCOMES:
Concordance of observed agreement using eSWAN and TOF images measured by Cohen's kappa coefficient | at inclusion
  Concordance of observed agreement for the detection of arterial occlusion between eSWAN and TOF images

SECONDARY OUTCOMES:
Concordance inter-observer agreement for the detection of arterial occlusion using eSWAN images measured by Cohen's kappa coefficient | at inclusion
  Concordance inter-observer agreement between the two readers for the detection of arterial occlusion using eSWAN images

CONTACTS AND LOCATIONS:
Overall Officials: Sebastien Verclytte, MD, Principal Investigator — GHICL